CLINICAL TRIAL: NCT05354570
Title: Phase II Study of Hemithoracic Intensity-Modulated Pleural Radiation Therapy (IMPRINT) for Patients With Pleural Metastases From Thymic Malignancies
Brief Title: A Study of Intensity-Modulated Pleural Radiation Therapy (IMPRINT) in People With Thymic Cancer That Has Spread to the Lining of the Lungs and Chest
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-098
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Thymic Malignancies; Pleural Metastases
Keywords: Intensity-Modulated Pleural Radiation Therapy (IMPRINT); 22-098

STUDY DESIGN:
Intervention Model Description: This is a single-arm Phase II single institution trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hemithoracic Intensity-Modulated Pleural Radiation Therapy (IMPRINT) (Experimental): Radiation will be administered over approximately 6 weeks to 50.4 Gy in 28 fractions with an optional SIB to gross residual disease.
  Interventions: Radiation: Intensity-Modulated Pleural Radiation Therapy (IMPRINT)

INTERVENTIONS:
Radiation: Intensity-Modulated Pleural Radiation Therapy (IMPRINT) — Radiation therapy will be administered over approximately 6 weeks at 50.4 Gy in 28 fractions, including an optional dose-painting SIB to gross residual disease up to 60 Gy while respecting normal tissue constraints.

SUMMARY:
The researchers are doing this study to find out whether hemithoracic intensity-modulated pleural radiation therapy (IMPRINT) is a safe treatment that causes few or mild side effects in people with pleural metastases from thymic malignancies. The researchers will also look at whether hemithoracic IMPRINT is effective against participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate on the study
* Patients must have a pathologically confirmed diagnosis of thymic malignancy. Thymic carcinoma is allowed.
* Patients must have radiologic or pathologic evidence of pleural metastases. Patients may have de novo stage IVA or recurrent disease in the pleura. Gross disease in the fissure is allowed if resected.
* No evidence of extrathoracic metastatic disease or contralateral pleural/pericardial disease.
* Patient age ≥ 18 years but ≤ 80 years at the time of consent
* Karnofsky performance status ≥ 80%
* Preoperative or Postoperative Pulmonary Function Tests: DLCO > 40% predicted (corrected for Hgb) and FEV1 ≥ 35% (corrected for Hgb)
* Glomerular filtration rate (GFR): ≥50 mL/min/1.73 m2 (must be calculated using estimated creatinine clearance (CrCl) by the Cockcroft-Gault (C-G) equation (Nephron 1976;16:31-41): CrCl (mL/min) = [140 - age (years)] x weight (kg) [x 0.85 for female patients] 72 x serum creatinine (mg / dL) ° In cases of concern about decreased renal function and potential high radiation dose to the kidneys, an optional nuclear medicine kidney function scan may be performed prior to radiation therapy to determine the functional contribution of each kidney.

Exclusion Criteria:

* Continuous oxygen use
* Patients with an acute flare of myasthenia gravis requiring addition of new medication in the past 6 months
* Prior nephrectomy on the contralateral side of the pleural metastases
* Prior thoracic radiation therapy preventing hemithoracic pleural IMRT. Prior thymic bed radiation is allowed. Prior pleural SBRT is allowed.
* Patients undergoing extrapleural pneumonectomy. Other surgical resection approaches of the pleural nodules (ex: P/D, debulking/metastasectomy) are allowed. Surgical resection of the primary thymic tumor is allowed.
* Acute congestive heart failure requiring hospitalization within the past 30 days.
* COPD requiring chronic oral steroid therapy of > 10 mg prednisone daily or equivalent at the time of registration. Inhaled corticosteroids are allowed
* Unstable angina requiring hospitalization and/or transmural myocardial infarction within the last 3 months
* History of interstitial lung disease
* Pregnant or lactating women
* Men or women not using effective contraception

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
assess the rate of radiation pneumonitis | 2 years
  as indicated by the rate of grade 3 or higher radiation pneumonitis defined by the NCI Common Terminology Criteria (CTC) version 5.0.

SECONDARY OUTCOMES:
progression-free survival (PFS) | 12 month
  PFS events will include death and/or progression of thymic malignancy due to local-regional or distant recurrence/progression. PFS will be calculated from the start of radiation treatment and will be estimated by the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Simone, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm